CLINICAL TRIAL: NCT04677699
Title: Combined Antibody Screening for Celiac and Diabetes Evaluation
Acronym: CASCADE
Status: Enrolling by invitation | Type: Observational
Sponsor: Pacific Northwest Research Institute (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Principal Investigator, William Hagopian, Director of Diabetes Program, Pacific Northwest Research Institute
Other Study IDs: WSIRB# 2020-078
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Type 1 Diabetes; Celiac Disease
Keywords: Type 1 Diabetes; Celiac Disease; Diabetes; Celiac; Gluten; Autoantibodies
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Celiac Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Birth Cohort: Newborns less than 8 months old and born in the state of Washington.
  Interventions: Diagnostic Test: Combined Risk Score
- Kids Cohort: Children ages 4-7 years and born in the state of Washington.
  Interventions: Diagnostic Test: Combined Risk Score

INTERVENTIONS:
Diagnostic Test: Combined Risk Score — Several factors will be analyzed to assign each subject combined risk score. This will assess the subject's risk of developing Type 1 Diabetes and/or Celiac Disease.

SUMMARY:
The CASCADE Study (Combined Antibody Screening for Celiac and Diabetes Evaluation) is an observational study whose primary goal is to show that population-based screening for advanced prediction of type 1 diabetes (T1D) and celiac disease (CD) is feasible to prevent diabetic ketoacidosis (DKA), improve celiac disease diagnosis, and ultimately gain public health acceptance to facilitate future prevention. It has two arms, a Birth Cohort and a Kids (cross sectional) Cohort.

ELIGIBILITY:
Inclusion Criteria:

* Child must be between 0 to 8 months in age or between 4 to 7 years in age. Child must be born in the state of Washington.

Exclusion Criteria:

-

Ages: 1 Day to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns and school aged children in the state of Washington.
Sampling Method: Non-Probability Sample
Enrollment: 64410 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Type 1 Diabetes | 5 years
Diagnosis of Celiac Disease | 5 years

SECONDARY OUTCOMES:
Severity of disease at diagnosis | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: William Hagopian, MD PhD, Principal Investigator — Pacific Northwest Research Institute
Locations (1):
- Pacific Northwest Research Institute, Seattle, Washington, United States